CLINICAL TRIAL: NCT05938751
Title: A Multicentric Mixed-methods Study About the Promotion of Self-determination in Young Adults With Autism: the TEAm_YOUNG ADULTS Program
Brief Title: An Intervention to Promote Self-determination in Young Adults With Autism: the TEAm_YOUNG ADULTS Program
Acronym: TEAm_YA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Collaborators: Hospital de Mataró (Other); Fundació Friends (Unknown); University of Barcelona (Other)
Responsible Party: Principal Investigator, Clara Andrés Gárriz, Principal Investigator, University Ramon Llull
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPCEE_TeamYoungAdults2020/2023
Record Dates: First submitted 2023-06-20; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Autism
Keywords: Self-determination; Intervention; Young adults; Mixed-methods
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Participants were assigned to the experimental group (which received the intervention) or to the control group (in a waiting list to receive the intervention after the conclusion of the study)
Masking Description: Masking was not possible due to the resources of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group received the TEAm_YOUNG ADULTS program, an intervention to promote and develop self-determination-related skills.
  Interventions: Behavioral: TEAm_YOUNG ADULTS program
- Waiting list group (No Intervention): Participants in this group were on the waiting list. That means they had to wait until the intervention group received the intervention and post-test evaluation to receive the intervention. They could keep their intervention as usual during the whole study.

INTERVENTIONS:
Behavioral: TEAm_YOUNG ADULTS program — The TEAm_YOUNG ADULTS program is an intervention to develop self-determination in young adults with autism. It consists of 20 1.5h weekly sessions. The intervention is conducted by two facilitators with expertise in autism and self-determination promotion. Groups are formed by 4 to 6 participants. The program can be applied online or in person. The first five sessions address specific characteristics and support needs of people with autism. The next ten sessions are focused on the development of self-determination. The last five sessions are focused on working with others and the closure of the group. The individual goals of every participant are considered in the beginning of the group and a weekly follow-up of goals is conducted.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to test the benefits of a program to develop self-determination in young adults with autism. Being self-determined means acting or causing things to happen in your life. It involves deciding, acting and believing in one-self.

The main question this clinical trial aims to answer is: Is the program developed useful to improve self-determination of young adults with autism?

Participants will receive a group intervention to support the development of their self-determination-related skills during 20 sessions (1 session/week).

Researchers will compare the self-determination outcomes between the group that receives the intervention and another group that is in a waiting list (and will receive the intervention later) to see if the changes are due to the intervention.

DETAILED DESCRIPTION:
This clinical trial employed a convergent mixed methods design. Quantitative and qualitative data were collected from the same participants and analyzed separately within a similar timeframe. The quantitative strand used self-reported and proxy-reported questionnaires to evaluate the impact of the TEAm_YOUNG ADULTS program on the self-determination of young adults with autism. The quantitative data was collected at baseline and at the completion of the program, after 5 months (20 sessions). In the qualitative strand, focus groups were used to explore changes in self-determination perceived by the participants that received the program and their acceptance of the intervention. The focus groups were conducted when finishing the group and after the self-reported questionnaires are answered. Proxy-reports were answered after the realization of the focus groups.

ELIGIBILITY:
Inclusion Criteria:

* To have a diagnosis of autism spectrum disorder in accordance with the criteria of the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), or of Asperger's syndrome, according to he DSM-IV
* To be between 17 and 30 years old.
* To have a verbal comprehension index higher than 70 in the Wechsler Adult Intelligence Scale-IV (WAIS-IV), to ensure a good comprehension of the program

Exclusion Criteria:

* Not having spoken language
* Having a condition that could significantly interfere in the group functioning, such as an acute psychotic disorder or challenging behavior

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Self-determination after 20 sessions (Quantitative measure: self-report) | At baseline and after the completion of the intervention (20 weeks later)
  Self-Determination Inventory: Student Report (SDI:SR). The Spanish adaptation was used.
  It is a self-report measure that evaluates the three dimensions of self-determination based on Causal Agency Theory (volitional action, agentic action and action-control beliefs) as well as the total self-determination scores.
Self-determination (Qualitative measure) | After the completion of the intervention (20 weeks later)
  Focus groups to evaluate the changes after the completion of the intervention. Questions related to the three dimensions of self-determination will be asked (volitional action, agentic action and action-control beliefs) in accordance with the quantitative measures to allow a joint display of the results following a mixed methodology (quantitative and qualitative). The focus groups will only be conducted for the intervention groups.
Change from baseline Self-determination after 20 sessions (Quantitative measure: proxy-report) | At baseline and after the completion of the intervention (20 weeks later)
  AUTODDIS Scale. It is a proxy-report measure that evaluates the three dimensions of self-determination based on Causal Agency Theory (volitional action, agentic action and action-control beliefs) as well as the total self-determination scores. The internal consistency of these sections was excellent (between α = .948 to α = .962), as well as for the entire scale (α = .983), and there is also evidence of its validity.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Andrés Gárriz, M.D., Principal Investigator — University Ramon Llull
Locations (2):
- Spain (2):
  - Ramon Llull University. Faculty of Psychology, Sciences of Education and Sports Blanquerna, Barcelona
  - University of Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andres-Garriz C, Farriols Hernando N, Gomez Hinojosa AM, Pretel-Luque T, Fabregues S, Mumbardo-Adam C. Promoting Self-Determination in Young Adults with Autism: A Multicenter, Mixed Methods Study. J Autism Dev Disord. 2025 Feb 15. doi: 10.1007/s10803-025-06739-6. Online ahead of print. PMID 39954217